CLINICAL TRIAL: NCT04785885
Title: Assessment of Clinical Onset of IV Heparin in Interventional Cardiology and Cardiac Surgery
Acronym: ACTPOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1651774
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Transcatheter Aortic Valve Replacement; Cardiac Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Transcatheter Aortic Valve Replacement: Patients receive 100U/Kg of IV heparin. An arterial sample activated clotting time (ACT) will be checked by iStat and hemochron
  Interventions: Diagnostic Test: iStat Handheld Blood Analyzer; Diagnostic Test: Hemochron
- Cardiac Valve Annuloplasty: Patients receive 300U/kg of IV heparin. An arterial sample activated clotting time (ACT) will be checked by iStat and hemochron
  Interventions: Diagnostic Test: iStat Handheld Blood Analyzer; Diagnostic Test: Hemochron

INTERVENTIONS:
Diagnostic Test: iStat Handheld Blood Analyzer — An easy-to-use blood analyzer that provides monitoring of heparin anticoagulation quickly for point-of-care testing. Testing will be done at baseline, 30s, 90s and 180s after heparin administration.
Diagnostic Test: Hemochron — An easy-to-use blood analyzer that provides monitoring of heparin anticoagulation quickly for point-of-care testing. Testing will be done at baseline, 30s, 90s and 180s after heparin administration.

SUMMARY:
The efficiency and promptness of heparin anticoagulation is necessary during the structural heart procedures to minimize time from insertion of cannulae to valve deployment in cardiac surgery. The goal of this study is to determine how rapidly the adequacy of heparin induced anticoagulation occurs using two different point of care activated clotting time technologies (iSTAT and Hemochron).

DETAILED DESCRIPTION:
Adequate anticoagulation is achieved in cardiac surgery and interventional cardiology procedures with intravenous (IV) administration of unfractionated heparin. The Activated clotting time (ACT) is routinely measured to assess adequacy of anticoagulation to prevent clotting/thrombotic complications from placement of foreign materials used during cardiac surgery and cardiology procedures. Alternative methods to measure adequacy of anticoagulation such as measurement of Anti-Xa level and Reaction (R) time as assessed by Thromboelastrography (TEG) have also been suggested. However, their use in clinical practice is limited by lack of Point of Care (POC) technology and need for additional expertise to run these tests.

The efficiency and promptness of heparin anticoagulation is necessary during the structural heart procedures to minimize time from insertion of cannulae to valve deployment in cardiac surgery. The time required to prevent major complications is on the order of seconds to minutes. The goal of this study is to determine how rapidly the adequacy of heparin induced anticoagulation occurs using two different point of care ACT technologies (iSTAT and Hemochron). It is hypothesized that anticoagulation can be determined by the iSTAT ACT device 30 seconds after administration of heparin. Measuring heparin effectiveness at 30 or 90 seconds instead of the usual 3-minute time period may allow for earlier cardiac intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients presenting for elective valvular surgery
* Interventional cardiology patients presenting elective Transcatheter Aortic Valve Replacement (TAVR)

Exclusion Criteria:

* Preoperative IV heparin administration within 12 hours of surgery
* Preoperative oral anticoagulant use within 24 hours of surgery
* Platelet count <120,000U/ml within 24 hours of surgery

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgical patients with intravenous (IV) administration of unfractionated heparin.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Activated Clotting Time (ACT) | Baseline, 30 seconds and 180 seconds after IV heparin administration
  Change in point of care activated clotting time (ACT) levels over time after IV heparin administration

SECONDARY OUTCOMES:
Laboratory-based anticoagulation | Baseline, 30 seconds and 180 seconds after IV heparin administration
  Laboratory-based anticoagulation measure of anti-Xa and TEG levels will be compared to point of care activated clotting time (ACT) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shyamal Asher, M.D., Principal Investigator — Rhode Island Hospital, Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falter F, MacDonald S, Matthews C, Kemna E, Canameres J, Besser M. Evaluation of Point-of-Care ACT Coagulometers and Anti-Xa Activity During Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2921-2927. doi: 10.1053/j.jvca.2020.06.027. Epub 2020 Jun 12. PMID 32620484
- [Background] Bolliger D, Tanaka KA. Point-of-Care Coagulation Testing in Cardiac Surgery. Semin Thromb Hemost. 2017 Jun;43(4):386-396. doi: 10.1055/s-0037-1599153. Epub 2017 Mar 30. PMID 28359133
- [Background] Heres EK, Speight K, Benckart D, Marquez J, Gravlee GP. The clinical onset of heparin is rapid. Anesth Analg. 2001 Jun;92(6):1391-5. doi: 10.1097/00000539-200106000-00006. PMID 11375810